CLINICAL TRIAL: NCT05058599
Title: Using a Reconstruction Technology With Facial Pathological Features to Auxiliary Diagnosis and Guarantee Patient Privacy
Brief Title: Reconstruction Technology to Auxiliary Diagnosis and Guarantee Patient Privacy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: 2021KYPJ77
Record Dates: First submitted 2021-09-16; First posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: 3D-reconstruction; Patient Privacy; Deep Learning; Digital Medicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- facial videos dataset: facial videos collected from Zhongshan Ophthalmic Center of Sun Yat-sen University.
  Interventions: Diagnostic Test: DM

INTERVENTIONS:
Diagnostic Test: DM — A new technology based on 3D reconstruction and deep learning algorithm to irreversibly erase the biometric attributes whilst retaining the clinical attributes needed for diagnosis and management

SUMMARY:
Medical data that contain facial images are particularly sensitive as they retain important personal biometric identity, privacy protection. We developed a novel technology called "Digital Mask" (DM), based on real-time three-dimensional (3D) reconstruction and deep learning algorithm, to extract disease-relevant features but remove patient identifiable features from facial images of patients.

ELIGIBILITY:
Inclusion Criteria:

* The quality of facial images should be clinically acceptable.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Outpatients from strabismus departments, paediatric ophthalmology departments, TAO departments, and ophthalmic plastic departments.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-05-10 (Actual); Primary Completion 2021-09-20 (Estimated); Study Completion 2022-01-30 (Estimated)

PRIMARY OUTCOMES:
Diagnostic consistency | baseline
  For each eye, both the diagnosis from the original videos and the diagnosis from the DM-reconstructed videos were recorded and compared. If the two diagnoses were consistent, it suggests that the reconstruction would be precise enough in clinical practice.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China